CLINICAL TRIAL: NCT06705803
Title: Prostate Ablation Registry and Database for Information, Surveillance, and Evaluation (PARADISE)
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 24-0111
Record Dates: First submitted 2024-11-14; First posted 2024-11-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Cancer Patients Undergoing Prostate Ablation: Patients with prostate cancer undergoing prostate ablation for the management of prostate cancer.
  Interventions: Procedure: Prostate Ablation

INTERVENTIONS:
Procedure: Prostate Ablation — Patients with prostate cancer undergoing prostate ablation for the management of prostate cancer.

SUMMARY:
Prostate cancer (PCa) is the most commonly diagnosed non-cutaneous cancer of men in the world. In 2023 alone, it is estimated that 288,300 US men will be diagnosed with prostate cancer and 34,700 will die from the disease despite the approval of multiple systemic agents. Due to advances in screening and imaging technology, PCa is now detected much earlier in its disease course. Prostate gland ablation for prostate cancer might provide the option for a "middle" ground between active surveillance (AS) and radical therapy by destroying prostate cancer in a minimally invasive or non-invasive fashion and thus limiting the morbidity. This treatment strategy is increasingly being offered to patients due to low morbidity but the data on long term oncologic efficacy and side effect profile is lacking for such a treatment strategy.

The purpose of this study is to create a database and prospective registry for data collection on patients with prostate cancer undergoing prostate ablation for the management of prostate cancer. Patients with biopsy-proven prostate cancer of any Gleason Grade will be entered into the registry as long as prostate ablation is used as the prostate cancer management modality. Historical data from 2017 to the present time will be added through chart review. Current and future patient data will be collected through chart review during the subject's clinical care. Only data available in the electronic medical record will be collected and no additional data will be collected for research purposes. No biospecimens will be collected, and there are no physical risks from study participation.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* ≥22 years of age
* Histologic diagnosis of prostate cancer
* Scheduled to undergo or have already undergone ablation of the prostate as part of routine clinical care or any ongoing clinical trials
* Prostate ablation performed with any of the following energy sources: cryotherapy, high-intensity focused ultrasound, irreversible electroporation, laser, microwave, radiofrequency ablation, or photodynamic therapy. Newer methods and instrumentation continue to be developed to ablate tissue, and these energy sources can be entered into the registry as clinical use begins

Exclusion Criteria:

* Under 21 Years of age.

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will collect data on all consecutive patients who have undergone prostate ablation at University of Chicago Medical Center without any exclusions. Patients will be consented at the UCMC campus as well as at River East.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with descriptive summarization of Prostate specific antigen (PSA) and its derivatives to represent clinicopathologic, interventions, and oncological outcomes | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Descriptive summarization of Prostate specific antigen (PSA) and its derivatives
Number of Participants with descriptive summarization of prostate biopsy | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Descriptive summarization of prostate biopsy to represent clinicopathologic, interventions, and oncological outcomes
Number of Participants with descriptive summarization of biomarkers | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Descriptive summarization of biomarkers to represent clinicopathologic, interventions, and oncological outcomes
Number of Participants with descriptive summarization of imaging findings | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Descriptive summarization of imaging findings to represent clinicopathologic, interventions, and oncological outcomes
Number of Participants with descriptive summarization of urination function | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Descriptive summarization of urination function to represent clinicopathologic, interventions, and genitourinary functional outcomes
Number of Participants with descriptive summarization of bowel function | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Descriptive summarization of bowel function to represent clinicopathologic, interventions, and genitourinary functional outcomes
Number of Participants with descriptive summarization of sexual function | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Descriptive summarization of sexual function to represent clinicopathologic, interventions, and genitourinary functional outcomes
Number of Participants with descriptive summarization of the overall quality of life parameters | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Descriptive summarization of the overall quality of life parameters to represent clinicopathologic, interventions, and genitourinary functional outcomes

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of prostate gland ablation in patients with localized prostate cancer measured on a continuous scale. | Follow up every 6 months (at minimum) for 2 years, and annually through 10 years of total follow-up after prostate cancer management.
  Data measured on a continuous scale will be expressed as a mean, standard deviation when normally distributed and as a median and interquartile range, when non-normally distributed.

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Sidana, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - The University of Chicago, Hyde Park, Illinois
  - The University of Cinncinatti, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided